CLINICAL TRIAL: NCT03921879
Title: A Phase 1 Study of OT-82 in Patients With Relapsed or Refractory Lymphoma
Brief Title: Safety and Efficacy of OT-82 in Participants With Relapsed or Refractory Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oncotartis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OT-82-001
Record Dates: First submitted 2019-03-12; First posted 2019-04-19 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, T-Cell; Lymphoma, Follicular; Lymphoma, Peripheral T-Cell; Lymphoma, Hodgkin
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, T-Cell; Lymphoma, Follicular; Lymphoma, T-Cell, Peripheral; Hodgkin Disease

STUDY DESIGN:
Intervention Model Description: Study OT-82-001 is a Phase 1, non-randomized, controlled, first-in-human, two stage (dose escalation and dose expansion) study evaluating multiple doses and schedules of orally administered OT-82 in patients with R/R lymphoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stage 1 Dose Escalation (Experimental): The dose escalation arm will use a modified 3+3 design to determine the maximum tolerated dose. or maximum tested dose.
  Interventions: Drug: OT-82 Dose Escalation
- Stage 2 Dose Expansion (Experimental): The dose expansion arm will use the maximum tolerated dose to determine preliminary efficacy.
  Interventions: Drug: OT-82 Dose Expansion

INTERVENTIONS:
Drug: OT-82 Dose Escalation — The starting OT-82 dose level will be16.5mg/m2 given orally as an oral suspension once daily on Days 1-3, 8-10, and 15-17 of each successive 28-day cycle. Dose escalation will follow a modified 3+3 design. There is no maximum duration of OT-82 treatment; however, treatment will be discontinued if there is unacceptable toxicity, disease progression, withdrawal of consent by the patient, noncompliance with study requirements, intercurrent illness, development of symptoms or conditions listed as exclusion criteria, or closure of the study by the Sponsor.
  Arms: Stage 1 Dose Escalation
Drug: OT-82 Dose Expansion — A total of 25 patients evaluable for disease response will be treated with OT-82 on Days 1-3, 8-10, and 15-17 of the 28-day cycle at the MTD or maximum tested dose determined from Stage 1. This may include patients treated at that dose in Stage 1 plus expansion at that dose during Stage 2. Evaluability for disease response requires that patients receive at least one dose of OT-82. There is no maximum duration of OT-82 treatment; however, treatment will be discontinued if there is unacceptable toxicity, disease progression, withdrawal of consent by the patient, noncompliance with study requirements, intercurrent illness, development of symptoms or conditions listed as exclusion criteria, or closure of the study by the Sponsor.
  Arms: Stage 2 Dose Expansion

SUMMARY:
This research study will test OT-82, which is an investigational ("research" or "experimental" ) drug. The study has two stages (Stage 1 and Stage 2). The purpose of Stage 1 is to determine the safety and tolerability and the maximum tolerated dose (MTD) or the maximum tested dose of OT-82 administered orally to participants. The purpose of Stage 2 is to determine the preliminary efficacy of OT-82 in relapsed or refractory lymphoma at the MTD or the maximum tested dose. Both parts of the study will also evaluate the pharmacokinetics (absorption, distribution, metabolism, elimination) of OT-82.

OT-82 treatment slowed the growth, reduced the size, or in some cases cured certain cancers in animal studies. It is hoped that participants with relapsed or refractory lymphoma treated with OT - 82 in this study will experience slowing tumor growth and/or reduction of tumor size.

DETAILED DESCRIPTION:
OT-82 affects an enzyme in the cancer cell called nicotinamide phosphoribosyltransferase (abbreviated NAMPT), which is involved with making energy for the cancer cell. OT-82 deprives the cancer cell of the energy that it needs to grow and divide.

This is a Phase 1, non-randomized (all participants will receive the study medication), open-label (identity of the study drug will be known to the participant and the study staff), controlled (the methods of the study are not random) study. Approximately 45 -50 participants at approximately 10 study centers across the USA will take part in this research study. The starting dose for Stage 1 is 16.5 mg/m2 per day. Participants in Stage 1 will be assigned a dose dependent on when he or she entered the study. Doses will increase for each new group of 3 to 6 participants until the maximum tolerated dose (MTD) or the maximum tested dose is reached. OT-82 is an oral liquid suspension that will be taken by mouth once per day for 3 days followed by a 4-day rest period.. A participant may continue to receive treatment with OT-82 as long as the study doctor feels it is in their best interest; as long as the participant does not develop intolerable side effects; as long as the participant wishes to remain in the study; or as long as the sponsor does not close the study.

Participants in Stage 2 of the study will receive either the MTD or the maximum tested dose of OT-82 determined in Stage 1. Assessment of anti-tumor activity will primarily focus on categorical objective response (Partial Response (PR) or Complete Response (CR)) as defined according to the consensus recommendations of the Lugano Classification criteria for malignant lymphoma (Cheson et al., 2014).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Provides signed informed consent before initiation of any study-specific procedures or treatment.
* Histologically (tumor tissue) confirmed diagnosis of lymphoma that has progressed despite prior treatment, and for which additional options leading to meaningful clinical benefit are not available. Lymphoma diagnoses may include the following:

  a. Confirmed histological diagnosis of the following types of B-cell Non-Hodgkin lymphoma (NHL): i. Low-grade B-cell NHLs including, but not limited to, FL, MCL, MZL, PMBL, LPC, or CLL/SLL. ii. Intermediate to high grade B-cell NHLs including, but not limited to DLBCL and other intermediate grade B-cell NHL, with disease progression following stem cell transplant or patient must be unwilling, unable or not an appropriate candidate for such. iii. Transformed Follicular Lymphoma. b. PTCL and others T-cell lymphoma, in which there is measurable non-cutaneous disease.

  c. Hodgkin's Lymphoma
* Measurable disease in all lymphoma classes except PTCL.

  1. Defined as nodal lesions >1.5 cm or extra-nodal, non-cutaneous lesions > 1.0 cm.
  2. Target lesions that have been previously irradiated and have not progressed since radiation are not considered measurable.
  3. Patients with PTCL may be eligible if they do not have measurable disease if they have skin disease.
* ECOG performance status of 0 or 1. This is a measure of a participant's ability to manage self care, mobility, work status, and other measures.
* Adequate baseline organ function.
* Adequate baseline hematologic (blood) function.
* Negative blood pregnancy test result obtained during screening if the patient is sexually mature woman who has not undergone a hysterectomy or ovary removal or has not been naturally postmenopausal for at least 24 consecutive months.
* Participant agrees to use acceptable contraceptive methods for the duration of time on the study, and continue to use acceptable contraceptive methods for 3 months after the last treatment with OT-82:
* Participant agrees to, and be capable of, adhering to the study visit schedule and other protocol requirements, including follow-up for survival.

Exclusion Criteria:

* Persistent clinically significant toxicities from previous anticancer therapy (excluding alopecia, which is permitted, and excluding Grades 2 and 3 laboratory abnormalities if they are not associated with symptoms, are not considered clinically significant by the Investigator, and can be managed with available medical therapies).
* Treatment with cytotoxic, biologic, or targeted therapies for lymphoma within 14 days before administration of the patient's first dose of OT-82.
* Treatment with an investigational drug within 28 days before administration of the patient's first dose of OT-82.
* Treatment with a stem cell transplant with an infusion of stem cells no less than 8 weeks before administration of the patient's first dose of OT-82. There should be no graft versus host disease > Grade 1 and participant should have discontinued all immunosuppressive therapy for such ≥ 2 weeks from OT-82 treatment.
* Radiation therapy within 14 days before administration of the patient's first dose of OT-82.
* Major surgical procedure within 28 days before administration of the patient's first dose of OT-82.
* Physical abnormality or medical condition that limits swallowing oral solutions, and/or has a history of non-adherence to oral therapies.
* Clinically significant gastrointestinal disorder that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Additional active malignancy that may confound the assessment of the study endpoints. If the participant has a past cancer history (i.e. active malignancy within 2 years before study entry) with substantial potential for recurrence, this must be discussed with the Sponsor before study enrollment. Patients with the following concomitant neoplastic diagnoses are eligible: nonmelanoma skin cancer and carcinoma in situ (including transitional cell carcinoma, cervical cancer, anal carcinoma, and melanoma in situ).
* Breastfeeding.
* Clinically significant cardiovascular disease including, but not limited to:

  1. Uncontrolled or any New York Heart Association Class III or IV congestive heart failure.
  2. Uncontrolled angina, history of myocardial infarction, unstable angina, or stroke within 6 months before study entry.
* Systolic blood pressure > 170 mm Hg or diastolic blood pressure > 110 mm Hg, or clinically significant arrhythmias not controlled by medication.
* Average QTc interval by QTcF on triplicate ECGs at screening or baseline > 470 msec (females) or > 450 msec (male).
* History of additional risk factors for a cardiac condition known as torsade de pointes (e.g., heart failure, low potassium, family history of long QT syndrome, use of concomitant medications that prolong the cardiac QT/QTc interval).
* Uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that, in the opinion of the Investigator, would put the patient at significant risk for pulmonary complications during the study (patient must not be dependent on oxygen).
* History of brain or leptomeningeal malignant disease (CNS imaging is not required before study entry unless there is a clinical suspicion of CNS involvement).
* Primary CNS lymphoma.
* Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days before administration of the patient's first dose of OT-82. Inhaled or topical steroids and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Uncontrolled illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known positive status for HIV and:

  1. Not receiving optimal anti-HIV therapy
  2. Demonstrated to be noncompliant with anti-HIV therapy.
  3. Has evidence of worsening HIV viral load (as assessed by HIV real-time qPCR).
  4. Not willing to attend HIV clinic follow-up at appropriate intervals.
* Active or chronic hepatitis B or hepatitis C (screening is not required).
* Any medical condition that, in the opinion of the Investigator, places the patient at unacceptably high risk for toxicity.
* Anticoagulation with warfarin or a direct thrombin inhibitor; a washout period of 7 days before administration of a patient's first dose of study drug is required for patients who are taken off these treatments (treatment with low molecular weight heparin is allowed).
* Requires a medication(s) that is a strong inhibitor of cytochrome CYP3A4 (boceprevir,clarithromycin, cobicistat, conivaptan, diltiazem, anoprevir/ritonavir, elvitegravir/ritonavir, grapefruit juice, idelasib, indinavir/ritonavir, itraconazole, ketoconazole, lopinavir/ritonavir, nefazodone, nelfinavir, paritaprevir/ritonavir/ombitasvir and/or dasabuvir, posaconazole, ritonavir, saquinavir/ritonavir, tipranavir/ritonavir, troleandomycin, voriconazole, and telithromycin).
* Requires a medication(s) that is a strong inducer of CYP3A4 (carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, and St John's wort).
* Requires a medication(s) that is a strong inhibitor of P-glycoprotein (P-gp) (amiodarone, carvedilol, clarithromycin, cyclosporine, dronedarone, elacridar, itraconazole, ketoconazole, lapatinib, lopinavir/ritonavir, propafenone, quinidine, ranolazine, reserpine, ritonavir, saquinavir/ritonavir, tacrolimus, telaprevir, tipranavir/ritonavir, verapamil).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Occurence of Dose Limiting Toxicities (DLT) in all participants during the Stage 1 Dose Escalation period | C1 (Days 1-28) through study completion.
  A DLT is a defined Adverse Events (AE) that limits the dosing schedule occurring during Cycle 1 regardless of Investigator attribution to OT-82.
Overall Response Rate in Participants with R/R Lymphoma | During Screening, at the end of Cycle 2 (C2) [each cycle is 28 days], then every 2 cycles thereafter until development of Progressive Disease (PD) up to week 24.
  Evaluation of antitumor response in patients with lymphoma will be by the Lugano Classification criteria for malignant lymphoma. Participant with undergo Computed Tomography (CT) scans or Magnetic Resonance Imaging (MRI) scans for participants unable to have CT imaging. Overall response is derived from time-point response assessments as follows:
  * CR: Complete disappearance of all detectible clinical evidence of disease and disease-related symptoms if present before therapy.
  * PR: Regression of measurable disease and no new sites.
  * SD: Failure to attain CR, PR, or PD.
  * PD: Any new lesion or increase by ≥50% of previously involved sites at nadir.
Response to OT-82 in Participants with Skin Involvement | Baseline (-14 days to -1 day before treatment), at the end of C1 and C2 (each cycle is 28 days), and every 2 cycles thereafter up to week 24.
  Assessments will be made using the modified Severity Weighted Assessment Tool (mSWAT) and will include skin biopsies and/or photographs as indicated.
Response to OT-82 in Participants with Bone Marrow Involvement | Baseline (-14 days to -1 day before treatment) and at week 24.
  Bone marrow studies will be performed to confirm CR in patients with known bone marrow involvement. Bone marrow aspirates (±biopsy) will be assessed.
Response to OT-82 in Participants with PTCL and known circulating clonal T lymphocytes | Baseline (-14 days to -1 day before treatment), at the end of C1 and C2 (each cycle is 28 days), and every 2 cycles thereafter up to week 24.
  Relevant clonal T cell populations will be measured from peripheral blood samples during treatment with OT-82 and compared to baseline measures.

SECONDARY OUTCOMES:
Evaluate the Maximum Plasma Concentration (Cmax) of OT-82 in Human Participants | Stage 1: Days 1,2,3,4,5,8,15,22, and 29; Stage 2: Days 1,2,8, and 15
  Blood samples taken prior to administration of the OT-82 dose will be assessed to determine the Cmax of OT-82 in human participants
Evaluate Time to Maximum Concentration (Tmax) of OT-82 in Human Participants | Stage 1: Days 1,2,3,4,5,8,15,22, and 29; Stage 2: Days 1,2,8, and 15
  Blood samples taken prior to administration of the OT-82 dose will be assessed to determine the Cmax of OT-82 in human participants
Evaluate the Area Under the Curve (AUC) of OT-82 in Human Participants | Stage 1: Days 1,2,3,4,5,8,15,22, and 29; Stage 2: Days 1,2,8, and 15
  Blood samples taken prior to administration of the OT-82 dose will be assessed to determine the AUC of OT-82 in human participants
Evaluate the Clearance (Cl) of OT-82 in Human Participants | Stage 1: Days 1,2,3,4,5,8,15,22, and 29; Stage 2: Days 1,2,8, and 15
  Blood samples taken prior to administration of the OT-82 dose will be assessed to determine the Clearance of OT-82 in human participants
Evaluate Visfatin Levels in Participants treated with OT-82 | Stage 1: Days 1,2,3,4,5,8,15,22, and 29; Stage 2: Days 1,2,8, and 15
  Visfatin, an enzyme involved in the mechanism of OT-82, will be measured with blood samples.

OTHER OUTCOMES:
Evaluate Tumor Tissue for Cancer Specific Genetic Mutations | Days 1-21 of Cycle 1 treatment
  Tumor tissue will be collected from the most recent archived tumor biopsy sample.
Evaluate Normal DNA Tissue | Baseline (-14 days to -1 day before treatment)
  Obtain DNA samples from the cheek of participants (buccal) to determine if genetic alterations are tumor-specific.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rowinsky, MD, Study Director — Oncotartis, Inc.
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No